CLINICAL TRIAL: NCT01348633
Title: Phase 1. Validation and Calibration Phase: Retinal Oxygen Saturation, Blood Flow, Vascular Function and High Resolution Morphometric Imaging in the Living Human Eye
Brief Title: Retinal Oxygen Saturation, Blood Flow, Vascular Function and High Resolution Morphometric Imaging in the Living Human Eye
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: Ontario Research Fund (Other)
Responsible Party: Principal Investigator, Chris Hudson, Professor, University of Toronto
Other Study IDs: ORF1
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Branch Retinal Artery Occlusion; Central Retinal Artery Occlusion; Branch Retinal Vein Occlusion; Central Retinal Vein Occlusion
Keywords: Doppler SD-OCT Blood Flow Technology; Retinal and choroidal blood flow; Canon Laser Blood Flowmeter
MeSH Terms: conditions — Retinal Artery Occlusion; Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Sub-study 1: The Quantitative, Doppler SD-OCT Blood Flow Technology will be validated and calibrated by manipulating end-tidal blood gases using the computer-controlled gas sequencer (Slessarev et al, 2005) in 15 healthy controls. Homeostatic inner retina blood flow values and the magnitude of vascular reactivity will be compared between Doppler SD-OCT blood flow technology and the Canon Laser Blood Flowmeter, an established standard, at specific locations within the retinal vascular tree.
- Sub-study 2: The Quantitative, Hyper-Spectral Imaging Derived Oxygen Saturation Maps of the major retinal vessels and capillary beds will be validated and calibrated in human volunteers using our novel and exact technique that allows the precise control of the partial pressure of oxygen (PO2) to induce controlled and safe levels of hypoxia. Oxygen saturation values will be compared to measured PO2 values (i.e. recognized standard) for various levels of hypoxia and will be used to provide in-sight into the properties of the data output e.g. effective operating range, linearity of response. At the end of the study, subjects will be returned to normoxic conditions to assess reproducibility of oxygen saturation maps.
- Sub-study 3: Subjects with symptoms of branch and central retinal artery and vein occlusion within the past 2 months will be used to validate the Doppler SD-OCT blood flow technology and the hyperspectral imaging derived oxygen saturation maps. In cases of central retinal vein and artery occlusion, imaging values (i.e. inner retinal and choroidal blood flow, oxygen saturation values of the major retinal vessels and the capillary beds of the retina and ONH) will be compared between the affected and unaffected eyes. In cases of branch occlusion, imaging values will be compared between the affected and unaffected quadrants of the affected eye and between the affected and unaffected eyes. The difference in inner retinal and choroidal blood flow for each eye will be calculated and compared between eyes.
- Sub-study 4: Calibration for retinal melanin, crystalline lens absorption, macular pigment, morphological variation and pre-retinal autofluorescence in healthy subjects (n=20 per decade, range 40 to 80yrs). Established reflectometric techniques to derive absorption values and autofluorescence techniques will be used to calculate correction values for each parameter that influences the hyper-spectral retinal and ON oxygen saturation imaging data (Keilhauer and Delori, 2006; Delori et al, 2007).
- Sub-study 5: Establishment of a database of healthy control imaging values (n=20 per decade, range 40 to 80yrs). A database of healthy control values will be established for each technology taking into account extraneous factors such as age (range 40 to 70 years) and gender. The healthy control database will be compared to the results of each individual patient in the prospective study phase of this proposed Research Program (see Prospective Study Phase, 3, Control group). Statistical confidence limits for abnormality at each time point, and for progression overtime, will be established. Measurements will be repeated at separate visits to establish repeatability.

SUMMARY:
Canadians fear loss of vision more than any other disability. Vision loss has an enormous impact on quality-of-life and is extremely costly from a societal and economic perspective. In 2001, more than 600,000 Canadians were estimated to have severe vision loss, accounting for 17% of total disability in Canada. One in 9 individuals experience severe vision loss by 65 years of age; however, this increases to 1 in 4 individuals by 75 years. The financial cost of vision loss in Canada is $15.8 billion per year. There is a general perception that vision loss is "normal with aging" but 75% of vision loss is estimated to be preventable. The major causes of severe vision loss are age-related macular degeneration (ARMD), glaucoma, particularly primary open-angle glaucoma (POAG), and diabetic retinopathy (DR). Canada is headed for an epidemic of age-related eye disease and, unless something is done to prepare for this, severe vision loss will have significant consequences in terms of societal and economic costs. Through this proposed Research Program, and in conjunction with our international academic and private sector partners, we will build and develop unique quantitative imaging technologies to permit non-invasive assessment of visual changes, structural changes in the thickness of the retina at the back of the eye and also changes in the amount of blood flowing through the blood vessels that feed the retina with oxygen. This research will add to our basic knowledge in predicting the development of sight-threatening change in patients with the three diseases, and facilitate earlier detection of the problem to help us discover earlier treatments for people with these conditions. The reliability of each imaging technology will be assessed by determining its ability to differentiate between diseased and healthy eyes. Cross-sectional analyses at yearly intervals, as well as change over time analyses, will be undertaken.

DETAILED DESCRIPTION:
There are a number of major steps that are required prior to the utilisation of these technologies in a clinical setting. This phase of the Proposal will aim to validate and calibrate the new technologies, explore the signal-to-noise ratio of RBF and oxygen saturation parameters, generate values to define the impact of absorption, morphological fundus variation and pre-retinal autofluorescence on oxygen saturation imaging and will establish a database of healthy control imaging values for both new technologies and the reproducibility of those measurements. Note: Sample size calculations have been conducted for all aspects of this phase of the protocol, based upon our extensive retinal vascular reactivity work. We will build and develop unique quantitative imaging technologies to that will permit us to explore the physiology of retinal and choroidal perfusion and vascular regulation, and retinal oxygenation.

Having completed the Validation and Calibration phase, this research will ultimately add to our basic knowledge in predicting the development of sight-threatening change in patients with the ARMD, diabetic retinopathy and primary open glaucoma, and facilitate earlier detection of the problem to help us discover earlier treatments for people with these conditions. The reliability of each imaging technology will be assessed by determining its ability to differentiate between diseased and healthy eyes. Through this proposed Research Program, we will build and develop unique quantitative imaging technologies to: Comprehensively assess the blood supply to, and vascular regulation characteristics of the posterior segment of the eye, a diagnostic capability that is currently severely limited. Assess oxygen saturation disturbances in the retina and ON that occur prior to clinically detectable changes, diagnostic capability that currently does not exist. Using the retinal blood supply and oxygen saturation parameters, we will derive net oxygen delivery to the retina and optic nerve head (ONH), a diagnostic capability that does not exist

ELIGIBILITY:
Inclusion Criteria:

* 20 to 80 years of age
* good vision in at least one eye (equivalent to 20/40 or better when wearing up-to-date spectacles)
* normal intraocular pressure (i.e. < 22 mm Hg)
* spectacle refraction between +/- 6.00 DS & / or +/- 2.50 DC

Exclusion Criteria:

* any ocular disease apart from retinal vein / artery occlusion (for stub study #3, patients with retinal vessel occlusion will be recruited)
* history of stroke, chronic lung disease (i.e. does not include seasonal asthma)
* taking medications with known effects on the blood vessels, other than medications to control blood glucose, blood pressure or cholesterol levels

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Flyers advertising the study will be posted on noticeboards within Toronto Western Hospital. The cohorts will be selected from the respondents to the flyer. Clincians in the Ophthalomology department in the Toronto Western Hopital will also offer the study to patients whom they consider to be potential participants.
Sampling Method: Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Validation and calibration of the Quantitative, Doppler SD-OCT Blood Flow Technology | 1 year
  Validation and calibration of the Doppler SD-OCT technology for their optimal utilisation in a clinical setting is required. We aim to explore the signal-to-noise ratio of retinal blood flow and oxygen saturation parameters, generate values to define the impact of absorption, morphological fundus variation and pre-retinal autofluorescence on oxygen saturation imaging and will establish a database of healthy control imaging values for both new technologies and the reproducibility of those measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Hudson, OD, PhD, Principal Investigator — University of Toronto, Toronto Western Research Institute, Toronto Western Hospital, University Health Network, University of Waterloo
Locations (1):
- Department of Ophthalmology and Vision Science, Toronto Western Research Institute, University Health Network, Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Tayyari F, Venkataraman ST, Gilmore ED, Wong T, Fisher J, Hudson C. The relationship between retinal vascular reactivity and arteriolar diameter in response to metabolic provocation. Invest Ophthalmol Vis Sci. 2009 Oct;50(10):4814-21. doi: 10.1167/iovs.09-3373. Epub 2009 Apr 1. PMID 19339742
- [Background] Keilhauer CN, Delori FC. Near-infrared autofluorescence imaging of the fundus: visualization of ocular melanin. Invest Ophthalmol Vis Sci. 2006 Aug;47(8):3556-64. doi: 10.1167/iovs.06-0122. PMID 16877429
- [Result] Slessarev M, Fisher JA, Volgyesi G, Prisman E, Mikulis D, Hudson C, Ansel C (2005). PATENT: A new method and apparatus to attain and maintain target end tidal gas concentrations (WO/2007/012170). International Application #: PCT/CA2005/001166. Filing Date: 28 / 07 / 2005. Pub Date: 01 / 02 / 2007.